CLINICAL TRIAL: NCT06118983
Title: Improving TRansitions ANd OutcomeS for Heart FailurE Patients in Home Health CaRe (I-TRANSFER-HF): A Type 1 Hybrid Effectiveness- Implementation Trial
Brief Title: Improving TRansitions ANd OutcomeS for Heart FailurE Patients in Home Health CaRe (I-TRANSFER-HF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Johns Hopkins University (Other); University of Colorado, Denver (Other); NYU Langone Health (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-06026204; R01HL169312 (NIH)
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
Keywords: home health care; hospital-to-home transition
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-TRANSFER-HF (Experimental): This is a 1-year long intervention period when I-TRANSFER-HF is in operation.
  Interventions: Other: I-TRANSFER-HF
- Standard of Care (usual care) (No Intervention): This is a baseline period of usual care (UC) with no intervention.

INTERVENTIONS:
Other: I-TRANSFER-HF — I-TRANSFER-HF is comprised of early and intensive HHC nurse visits and an outpatient visit within 7 days of discharge. Using a Hybrid Type 1, stepped wedge randomized trial design, we will test the effectiveness and implementation of I-TRANSFER-HF in partnership with 4 geographically diverse dyads of hospitals and HHC agencies ("hospital-HHC agency" dyads) across the US.
  Arms: I-TRANSFER-HF

SUMMARY:
This study is trying to improve the hospital-to-home transition for people with heart failure who receive home care services. The study will test an intervention called I-TRANSFER-HF, which differs from usual care by combining early home health nurse visits and outpatient medical appointments.

The study is interested in two questions:

1. Is I-TRANSFER-HF better than usual care at preventing heart failure patients from returning to the hospital within 30 days?
2. Are there parts of I-TRANSFER-HF that are easy or hard to implement in the real world?

The researchers will answer these questions by testing the intervention among pairs of hospitals and home health agencies across the country. During the study, the hospital-agency pairs will be asked to implement I-TRANSFER-HF. The researchers will then compare the results from before and after I-TRANSFER-HF was adopted. They will also interview people from these hospitals and agencies to see how I-TRANSFER-HF is being implemented under real-world conditions.

DETAILED DESCRIPTION:
The investigators' will test two hypotheses:

Hypothesis 1 (H1): Compared to usual care, adults with heart failure who receive the I-TRANSFER-HF intervention will have fewer 30-day readmissions, ED visits, and greater days at home. The four hospital-agency pairs will all begin the study with a baseline period of no intervention and then randomly selected to start the intervention phase at different points in time. Medicare claims data from each hospital-agency pair will be used to determine outcomes, and these data will be supplemented with national claims data for external controls not in the study to test the effectiveness of the I-TRANSFER-HF intervention.

Hypothesis 2 (H2): Compared to usual care, heart failure patients who receive I-TRANSFER-HF will have a higher proportion of timely first week HHC nursing visits (within 2 days of hospital discharge, plus 2 more) and outpatient visits (within 7-days of discharge). Given the rise of telemedicine, the study will test the association between the type of outpatient visit (in-person vs. virtual), its timing, and its association with outcomes. H2 requires conducting qualitative interviews with key stakeholders across the 4 hospital-agency pairs to identify barriers and facilitators that influence I-TRANSFER-HF's implementation. The study will assess the intervention's acceptability, feasibility, fidelity, and adaptation with interviews and Medicare claims data using a multi-methods approach and guided by the updated Consolidated Framework for Implementation Research (CFIR 2.0).

ELIGIBILITY:
Aim 1, Inclusion Criteria:

* Adults hospitalized for HF who transition from participating hospitals to their partner HHC agency during the study period.

Aim 1, Exclusion Criteria:

* Patients hospitalized for HF and discharged: home without HHC, or to an inpatient rehabilitation facility, skilled nursing facility, or hospice; patients with end stage renal disease on dialysis and those with left ventricular devices.

Aim 2, Inclusion Criteria:

- Healthcare professional involved in the transition of heart failure patients from the acute care setting (hospital) to HHC (home health care) agencies, and the implementation of the I-TRANSFER-HF at one of the four participating hospital-HHC dyads.

Aim 2, Exclusion Criteria:

- Healthcare professional not involved in the transition of heart failure patients from the acute care setting (hospital) to HHC (home health care) agencies, and the implementation of the I-TRANSFER-HF at one of the four participating hospital-HHC dyads.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1094 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
All-cause 30-day hospital readmission | 30 days following post-Index HF Hospitalization
  All-cause 30-day hospital readmission among adults hospitalized for heart failure who receive home health care after discharge and receive the I-TRANSFER-HF protocol compared to usual care, as assessed by Medicare claims
Number of Eligible patients | 12 months
  Number of heart failure patients eligible to receive I-TRANSFER-HF as assessed by Medicare claims data
Number of Eligible Patients Who Received Protocol Components | 12 months
  Number of heart failure patients who received both components of I-TRANSFER-HF (front-loaded home health nurse visits and early outpatient medical follow-up), one, or none as assessed by Medicare claims data
Modality of outpatient follow-up | 12 months
  The modality of outpatient follow-up received (in-person vs. virtual visit) as assessed by Medicare claims data
Timeliness of Post-Hospital Discharge Home Health Nursing Evaluation | 12 months
  The timeliness of first-week nursing visits within 2 days of hospital discharge as assessed by Medicare claims data
Timeliness of Post-Hospital Outpatient Follow-Up | 12 months
  The timeliness of outpatient visits within 7 days of hospital discharge as assessed by Medicare claims data
Feasibility of implementing I-TRANSFER-HF (Qualitative Interviews) | 30 days after intervention (year of intervention)
  Feasibility will be assessed through qualitative interviews with site stakeholders
Feasibility of implementing I-TRANSFER-HF (Surveys) | 30 days after intervention (year of intervention)
  Feasibility will be measured through the completion of the validated, 4-item, Feasibility of Intervention Measure (FIM). Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). The score is calculated as the mean. The scale for this measure ranges from 4-20 with higher scores indicating greater perceived feasibility of the intervention.

SECONDARY OUTCOMES:
All-cause 30-day ED visits | 30 days following post-Index heart failure Hospitalization.
  All-cause 30-day emergency department visits among adults hospitalized for heart failure who receive home health care after discharge and receive the I-TRANSFER-HF protocol compared to usual care, as assessed by Medicare claims data
Days at home among adults hospitalized for heart failure who receive home health care after discharge and receive the I-TRANSFER-HF protocol compared to usual care, as assessed by Medicare claims | During a 12-month period (year of intervention)
  Days at home will be calculated as 365 days minus the number of inpatient days in an acute care facility, an inpatient rehabilitation facility, a skilled nursing facility, or an inpatient hospice unit.
Acceptability of I-TRANSFER-HF - Qualitative Interviews | 30 days after intervention (year of intervention)
  Acceptability will be assessed through qualitative interviews.
Acceptability of Intervention Measure for the I-TRANSFER-HF Study - Survey | 30 days after intervention (year of intervention)
  Acceptability will be assessed through the 4-item, validated, Acceptability of Intervention Measure (AIM). Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). The score is calculated as the mean. The scale for this measure ranges from 4-20 with higher scores indicating greater perceived acceptability of the intervention.
Fidelity of I-TRANSFER-HF (Participant-Completed) | 30 days after intervention (year of intervention)
  Fidelity will be assessed by extent to which I-TRANSFER-HF is implemented by the study site teams. Fidelity will be measured using participant-completed fidelity checklists. These checklists will be developed during the implementation process.
Fidelity of I-TRANSFER-HF (Observational Ratings) | 30 days after intervention (year of intervention)
  Fidelity will be assessed by extent to which I-TRANSFER-HF is implemented by the study site teams. Fidelity will be measured using observational fidelity ratings conducted by site champions. These checklists will be developed during the implementation process.
Adaptation of I-TRANSFER-HF | 30 days after intervention (year of intervention)
  Adaptation will be assessed with qualitative interviews to document how the intervention was modified and refined during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Madeline R Sterling, MD, MPH, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - VNS Health Partners in Care, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sterling MR, Espinosa CG, Spertus D, Shum M, McDonald MV, Ryvicker MB, Barron Y, Tobin JN, Kern LM, Safford MM, Banerjee S, Goyal P, Ringel JB, Rajan M, Arbaje AI, Jones CD, Dodson JA, Cene C, Bowles KH. Improving TRansitions ANd outcomeS for heart FailurE patients in home health CaRe (I-TRANSFER-HF): a type 1 hybrid effectiveness-implementation trial: study protocol. BMC Health Serv Res. 2024 Oct 1;24(1):1160. doi: 10.1186/s12913-024-11584-x. PMID 39354472